CLINICAL TRIAL: NCT06294015
Title: Efficacy of 20% Autologous Serum Drops in the Treatment of Corneal Epitheliopathy Associated With Antihypertensive Glaucoma Drops.
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-5009
Record Dates: First submitted 2024-01-31; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Corneal Epitheliopathy; Glaucoma; Corneal Disease; Dry Eye
MeSH Terms: conditions — Glaucoma; Corneal Diseases; Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 20% Autologous serum eye drops + Artificial tear drops (Experimental)
  Interventions: Biological: 20% ASED + AT
- 0.9% NS eye drops + Artificial tear drops (Placebo Comparator)
  Interventions: Drug: 0.9% NS + AT

INTERVENTIONS:
Biological: 20% ASED + AT — Participants receive 20% Autologous Serum Eye Drops prepared by the hospital laboratory from the patients blood, diluted with sterile 0.9% sodium chloride to achieve the desired concentration. These drops are administered 6 times daily in one eye for two months. On top of this intervention is standard artificial tears therapy (Refresh Plus), applied four times daily.
  Arms: 20% Autologous serum eye drops + Artificial tear drops
Drug: 0.9% NS + AT — Participants in the placebo group receive eye drops consisting of sterile 0.9% sodium chloride solution, which serves as the placebo. The placebo solution is administered 6 times daily in one eye for two months. Alongside the placebo drops, participants continue with standard artificial tears therapy (Refresh Plus), applied four times daily throughout the study duration.
  Arms: 0.9% NS eye drops + Artificial tear drops

SUMMARY:
Introduction: Glaucoma is the second leading cause of blindness globally. Most anti-hypertensive drops contain preservatives harmful to the corneal epithelium, with up to 78% of treated patients reporting dry eye symptoms. Autologous serum eye drops (ASED), contains essential growth factors and nutrients which may promote corneal and conjunctival integrity, offering benefits over traditional treatments. This study investigates the efficacy of 20% ASED over placebo in the treatment of corneal epitheliopathies in patients with glaucoma treated with antihypertensive drops.

Methods: The present study is a triple-blinded, randomized controlled trial that anticipates to enroll 25 patients (50 eyes) with bilateral corneal epitheliopathy secondary to antihypertensive glaucoma treatments. Patients will receive autologous serum eye drops in one eye and placebo in the contralateral eye for two months, in addition to standard artificial tears treatment.

The primary outcome is the comparison of National Eye Institute (NEI) scores between autologous serum drops and placebo-treated eyes at two months. Secondary outcomes include Schirmer's test scores, visual acuity, tear break-up time (TBUT), Ocular Surface Disease Index (OSDI) scores, intraocular pressure, and complication rates.

The study aims to analyze the effectiveness of autologous serum eye drops in treating corneal epitheliopathies in glaucoma patients, potentially offering a new therapeutic avenue.

ELIGIBILITY:
Inclusion Criteria:

* Patients with glaucoma who developed corneal epitheliopathy secondary to antihypertensive drops;
* Epitheliopathy refractory to conventional therapies (Artificial Tears, ointment, topical cyclosporine or punctal plug, etc.);
* National Eye Institute score of 3 or more for both eyes;
* Adults aged 18 to 90 years inclusively.

Exclusion Criteria:

* Corneal epitheliopathy of other origin (ie. mechanical, neurotrophic, toxic, post-infectious, limbal stem cell deficiency);
* Glaucoma surgery within the last six (6) months;
* Previous corneal surgery;
* Active autoimmune disease;
* Frequent contact lense wear;
* Pregnant or actively breast-feeding;
* Known systemic infection with HIV, hepatitis B and C or syphilis;
* Known severe anemia (Hb < 100 g/L);
* Inability to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
National Eye Index Scores | 2 months
  Compare NEI scores at 2 months between eyes treated with ASED 20% versus placebo in patients with corneal epitheliopathy secondary to antihypertensive glaucoma treatments.

SECONDARY OUTCOMES:
Schirmer Test | 2 months
  Compare Schirmer Test scores at 2 months between eyes treated with ASED 20% versus placebo in patients with corneal epitheliopathy secondary to antihypertensive glaucoma treatments.
Visual Acuity | 2 months
  Compare visual acuity at 2 months between eyes treated with ASED 20% versus placebo in patients with corneal epitheliopathy secondary to antihypertensive glaucoma treatments.
Tear Break Up Time | 2 months
  Compare tear break up time at 2 months between eyes treated with ASED 20% versus placebo in patients with corneal epitheliopathy secondary to antihypertensive glaucoma treatments.
Ocular Surface Disease Index | 2 months
  Compare ocular surface disease index scores at 2 months between eyes treated with ASED 20% versus placebo in patients with corneal epitheliopathy secondary to antihypertensive glaucoma treatments.
Intraocular Pressure | 2 months
  Compare intraocular pressure at 2 months between eyes treated with ASED 20% versus placebo in patients with corneal epitheliopathy secondary to antihypertensive glaucoma treatments.
Complication rates | 2 months
  Compare complications at 2 months between eyes treated with ASED 20% versus placebo in patients with corneal epitheliopathy secondary to antihypertensive glaucoma treatments.